CLINICAL TRIAL: NCT01829126
Title: Development and Prevention of Severe Heart Disease in Systemic Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gabriele Valentini (Other)
Collaborators: European Union (Other); University of Giessen (Other); University of Zurich (Other); University of Paris 5 - Rene Descartes (Other); University of Florence (Other); University of Basel (Other); University College, London (Other); Charite University, Berlin, Germany (Other); University of Pecs (Other); University of Leeds (Other); Schoen Klinik Hamburg Eilbek (Other)
Responsible Party: Sponsor-Investigator, Gabriele Valentini, Prof. Gabriele Valentini, University of Campania Luigi Vanvitelli
Organization: University of Campania Luigi Vanvitelli (Other)
Other Study IDs: HEALTH-F5-2012-305495-OT5
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Systemic Sclerosis; Cardiac Diseases; Heart Block; Cardiac Arrhythmia; Congestive Heart Failure
MeSH Terms: conditions — Scleroderma, Systemic; Heart Diseases; Heart Block; Arrhythmias, Cardiac; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- CCB: Patients receiving calcium channel blockers (CCB)
- ACEi: Patients receiving angiotensin converting enzyme inhibitors (ACEi)
- CCB and ACEi: Patients receiving calcium channel blockers (CCB) and angiotensin converting enzyme inhibitors (ACEi)
- No treatment: Patients not receiving calcium channel blockers (CCB) and/or angiotensin converting enzyme inhibitors (ACEi)

SUMMARY:
Systemic sclerosis is an orphan, multiorgan disease affecting the connective tissue of the skin and all internal organs. Cardiac involvement, mainly characterised by small intramyocardial coronary artery involvement and myocardial fibrosis, can cause the development of impaired diastolic ventricular filling, cardiac blocks and ventricular arrhythmias, and can ensue in congestive heart failure and sudden death. Until now, no drug has been proven to have a therapeutic effect on SSc myocardial disease on an evidence-based level. Short-term trials and retrospective studies have suggested a favourable and protective effect of calcium channel blockers and angiotensin converting enzyme inhibitors in patients with myocardial involvement. However, no data are presently available on the prevention and treatment of severe heart disease.

This observational trial is part of the collaborative project "DeSScipher", one out of five observational trials to decipher the optimal management of systemic sclerosis. Aim of this observational trial is to assess the efficacy and safety of calcium channel blockers and angiotensin converting enzyme inhibitors in asymptomatic SSc patients with cardiac involvement.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile and adult systemic sclerosis patients, with diagnosis according to the SSc ACR/EULAR criteria or the PRES/ACR/EULAR juvenile SSc criteria respectively
* Asymptomatic (for cardiac disease) systemic sclerosis patients at risk for severe heart disease with at least one of the following risk factors: male sex and/or DLCO lower than 80% and/or sPAP > 30 mmHg and/or synovitis and/or joint contractures and/or digital ulcers and/or proteinuria.

Asymptomatic for cardiac disease is defined by patients without dyspnea NYHA >/= II, without palpitations and without bilateral leg edema.

Exclusion Criteria:

* Any significant pulmonary parenchymal (FVC < 70% and/or DLCO < 70%), pulmonary vascular (estimated systolic PAP > 40 mmHg), gastrointestinal (malabsorption syndrome or paralytic ileus) or renal (serum creatinine level >1.2 mg/dl, dialysis or previous scleroderma renal crisis) involvement
* Patients with dyspnea class NYHA >/= II
* Patients with palpitations
* Patients with bilateral leg edema.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population are adult and juvenile SSc patients from the EUSTAR cohort (MEDSonline database) and the jSScWG cohort
Sampling Method: Probability Sample
Enrollment: 765 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of CB, VA, pacemaker implantation, congestive heart failure and sudden death | 1 years
  Cumulative incidence of cardiac blocks, ventricular arrhythmias, pacemaker implantation, congestive heart failure and sudden death.

OTHER OUTCOMES:
Incidence of drug-related adverse events, incidence of withdrawal from treatment due to drug-related adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Müller-Ladner, Prof., Study Chair — Justus-Liebig-University Gießen, Kerckhoff Clinic, Departement of Rheumatology and Clinical Immunology; Gabriele Valentini, Prof., Principal Investigator — Policlinico, Via Pansini, Napoli-Italia
Locations (11):
- Université Paris Descartes, Hôpital Cochin, Service de Rhumatologie A & INSERM 1016, Paris, France
- Germany (3):
  - Justus-Liebig-University Gießen, Kerckhoff Clinic, Departement of Rheumatology and Clinical Immunology, Bad Nauheim
  - Charité Universitätsmedizin Berlin, Charité Centrum 12 für Innere Medizin und Dermatologie, Medizinische Klinik mit Schwerpunkt Rheumatologie und Klinische Immunologie, Berlin
  - Centre for Pediatric Rheumatology, Klinikum Eilbek, Hamburg
- Pecsi Tudomanyegyetem - University of Pecs, Pécs, Hungary
- Italy (2):
  - University of Florence, Denothe Centre, Division of Rheumatology AOUC, Department of Biomedicine, Florence
  - Policlinico, Via Pansini, Napoli-Italia
- Switzerland (2):
  - Felix-Platter Spital, University of Basel, Basel
  - University of Zurich, Department of Rheumatology, Zurich
- United Kingdom (2):
  - The Universitiy of Leeds, Division of Rheumatic and Musculoskeletal Disease, St James's University Hospital, Leeds
  - Royal Free Hospital, University College London, London